CLINICAL TRIAL: NCT05560542
Title: Prophylactic Efficacy and Safety of Intrathecal Dexamethasone, Atropine or Their Combination on Morphine Induced Post-operative Nausea and Vomiting on Patients Undergoing Caesarean Section With Spinal Anaesthesia
Brief Title: Intrathecal Dexamethasone and Atropine on Morphine Induced Post-operative Nausea and Vomiting on Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Shaban Abd Elbadea Khalifa, Anaesthesia and ICU Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAD-PONV-SCS
Record Dates: First submitted 2022-09-17; First posted 2022-09-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Morphine Adverse Reaction
MeSH Terms: interventions — Atropine; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone group (D) (Other): Patients will receive intrathecal hyperbaric bupivacaine 0.5% in a dose of 12.5 mg (2.5 ml) mixed with morphine in a dose of 200 µg (0.5 ml was withdrawn from a syringe containing 4 mg morphine sulfate diluted in 10 ml normal saline) [Total volume 4 ml], followed by intrathecal dexamethasone 4 mg (1ml).
  Interventions: Drug: Atropine and Dexamethasone
- Atropine group (A) (Other): Patients will receive intrathecal hyperbaric bupivacaine 12.5 mg (2.5 ml 0.5%) mixed with morphine 200 µg (0.5 ml) and atropine100 µg (0.5 ml was withdrawn from a syringe containing 2 mg atropine sulfate diluted in 10 ml normal saline) [Total volume 3.5 ml].
  Interventions: Drug: Atropine and Dexamethasone
- Dexamethasone and Atropine group (DA) (Other): Patients will receive intrathecal hyperbaric bupivacaine in a dose of 12.5 mg (2.5 ml) mixed with morphine 200 µg (0.5 ml) and atropine 100 µg (0.5 ml), followed by intrathecal injection of dexamethasone 4 mg (1 ml) [Total volume 4.5 ml] .
  Interventions: Drug: Atropine and Dexamethasone

INTERVENTIONS:
Drug: Atropine and Dexamethasone — Intrathecal dexamethasone, atropine or their combination.

SUMMARY:
Pain is a major problem during the postoperative period and can be considered as a challenge for the anesthesiologist. Low dose intrathecal morphine is proven efficient as a mode to reduce postoperative pain. Morphine has many complications like post-operative nausea and vomiting (PONV). the investigators will investigate the utility of intrathecal (IT) atropine and dexamethasone for prevention of morphine induced PONV as a primary outcome in parturient undergoing CS under spinal bupivacaine anesthesia plus morphine sulfate as an adjuvant.

DETAILED DESCRIPTION:
Pain is a major problem during the postoperative period and can be considered as a challenge for the anesthesiologist. Low dose intrathecal morphine is proven efficient as a mode to reduce postoperative pain in many surgical areas including Caesarean delivery. Morphine has many complications namely pruritus, and post-operative nausea and vomiting (PONV). The other risk factors for the development of PONV include female gender, non-smoker status, general anesthesia with inhalational anesthetics and surgical factors (duration and type of surgery). The supplementation of morphine, however raises the occurrences of postoperative nausea and vomiting (PONV) in these patient To tackle this problem, the investigators have to use the combination therapy of antiemetics like a serotonin receptor antagonist of either intravenous (IV) ondansetron or granisetron with IV dexamethasone is administered after the administration of intrathecal morphine. Dopamine receptor antagonists e.g. droperidol and metoclopramide are commonly used, but they carry the risk of extrapyramidal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18-45 years old
3. ASA: 1, 2
4. Elective caesarean section under spinal anaesthesia.

Exclusion Criteria:

1. Patient refusal.
2. Contraindications to spinal anaesthesia as coagulopathy, infection at site of injection, hemodynamic instability and uncooperative patient.
3. Contraindications to administration of morphine as asthmatic patient and hypersensitivity and contraindications to any of the study drugs.
4. Adult-Emergency CS as there is no time for preparation and risk on fetus and mother for time consuming

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult Pregnant Female
Enrollment: 150 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of PONV | 24 hour
  Incidence and severity of PONV by designing questionnaire and specific scale:
  1. no nausea or vomiting
  2. mild nausea and vomiting but no need to treatment
  3. moderate nausea and vomiting that need treatment
  4. severe form of nausea and vomiting and resistant to treatment

SECONDARY OUTCOMES:
Antiemetic | 24 hour
  Total dose of post-operative rescue antiemetic (ondansetron in mg) for 24 hour
Post-operative pain profile | 24 hour
  Post-operative visual analog scale (1: no pain and 10: the most severe experienced pain ) for 24 hour.
Incidence of Side Effects | 24 hour
  Anticipated side effects as shivering and hypotension( number of patients and severity)
Analgesia | 24 hour
  Time to the first post-operative rescue analgesic for 24 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Araujo R; PAMA Trial. [Pain Management, Local Infection, Satisfaction, Adverse Effects and Residual Pain after Major Open Abdominal Surgery: Epidural versus Continuous Wound Infusion (PAMA Trial)]. Acta Med Port. 2017 Oct 31;30(10):683-690. doi: 10.20344/amp.8600. Epub 2017 Oct 31. Portuguese. PMID 29268061
- [Background] Gwirtz KH, Young JV, Byers RS, Alley C, Levin K, Walker SG, Stoelting RK. The safety and efficacy of intrathecal opioid analgesia for acute postoperative pain: seven years' experience with 5969 surgical patients at Indiana University Hospital. Anesth Analg. 1999 Mar;88(3):599-604. doi: 10.1097/00000539-199903000-00026. PMID 10072014
- [Background] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Background] Rusch D, Eberhart LH, Wallenborn J, Kranke P. Nausea and vomiting after surgery under general anesthesia: an evidence-based review concerning risk assessment, prevention, and treatment. Dtsch Arztebl Int. 2010 Oct;107(42):733-41. doi: 10.3238/arztebl.2010.0733. Epub 2010 Oct 22. PMID 21079721
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Wang JJ, Ho ST, Lee SC, Liu YC, Liu YH, Liao YC. The prophylactic effect of dexamethasone on postoperative nausea and vomiting in women undergoing thyroidectomy: a comparison of droperidol with saline. Anesth Analg. 1999 Jul;89(1):200-3. doi: 10.1097/00000539-199907000-00036. PMID 10389804